CLINICAL TRIAL: NCT01625962
Title: Brain Indices of Risk for Posttraumatic Stress Disorder After Mild Traumatic Brain Injury
Brief Title: Brain Indices of Risk for Posttraumatic Stress Disorder (PTSD) After Mild Traumatic Brain Injury (mTBI)
Status: Completed | Type: Observational
Sponsor: INTRuST, Post-Traumatic Stress Disorder - Traumatic Brain Injury Clinical Consortium (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: INTRuST-BRI
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2015-08

CONDITIONS: PTSD
Keywords: PTSD; mTBI; mild TBI; extracranial injury; ECI; Brain Indices
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- mTBI: Service members who have sustained "impact-induced mTBI" or "blast-induced mTBI" (n = 74 completers)
- ECI: Service members who have sustained an extracranial injury (ECI) with no evidence of TBI (n = 32 completers)

SUMMARY:
This is a prospective, longitudinal cohort study to evaluate the associations between indices of brain structure and function (measured at baseline, as soon as possible after injury) and course of post-traumatic stress disorder (PTSD) symptoms. Subjects will be service members who have sustained mild traumatic brain injury (classified as either "impact-induced mTBI" or "blast-induced mTBI"; n = 100 completers) or an extracranial injury (ECI) with no evidence of traumatic brain injury (TBI) (n = 100 completers). Subjects will complete an assessment battery at baseline and 6 months later that includes (1) structural magnetic resonance imaging (MRI) and diffusion tensor imaging (DTI) derived from a 3-Tesla magnet; (2) event-related brain potentials (ERPs) derived from brain electrical activity; (3) neurocognitive tests; and (4) neurological soft signs (NSS). Specific indices of brain structure and function derived from these assessments are hypothesized to demonstrate a significant relationship with course of PTSD symptoms, which will be measured at baseline, 3 months, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Injured while deployed or stateside
2. Must be diagnosed TBI positive or certified as TBI negative by a licensed medical practitioner using Department of Defense (DoD) criteria
3. For mTBI subjects, an initial score of 13-15 on the Glasgow Coma Scale
4. Aged 18-50
5. Defense Enrollment Eligibility Reporting System (DEERS) eligible

Exclusion Criteria:

1. Unable or unwilling to provide informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization ("unable" includes cases in which the potential subject cannot read and understand English well enough to provide informed consent)
2. Penetrating head injury
3. Medical chart reveals a history of significant neurological condition(s) (reviewed on a case by case basis)
4. Diagnosis with or undergoing treatment for an illness that could affect brain function (reviewed on a case-by-case basis)
5. History of major psychiatric condition(s) that interfere with daily functioning as revealed in the medical chart or by the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID)
6. Record of drug or alcohol abuse or dependence in the past six months as documented in medical history review
7. Medical chart or SCID reveals current or lifetime PTSD diagnosis related to non-combat life events that occurred prior to most recent deployment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Service members who have sustained mild TBI or extracranial injury (ECI), and have received care at Walter Reed National Military Medical Center or Fort Belvoir Community Hospital.
Sampling Method: Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2011-10; Primary Completion 2015-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Correlation between brain structure and function and PTSD symptoms, as measured by the Clinician-Administered PTSD Scale (CAPS) | Change between Baseline and 3-months and 6-months
  To evaluate the associations between (1) baseline indices of brain structure and function and (2) course of PTSD symptoms in service members with TBI and ECI over the 6-month follow-up period.

SECONDARY OUTCOMES:
Correlation between brain structure and function and cognitive, functional, headache, behavioral and quality of life measures | Change between Baseline and 3-months and 6-months
  To evaluate the associations between (1) the selected baseline indices of brain structure and function, and (2) course of post-concussive symptoms, self-reported health status, including headache, overall emotional distress, and quality of life over the 6-month follow-up period.
Evaluate effect of injury type and brain structure and function | Change between Baseline and 3-months and 6-months
  To evaluate the effect of type of injury (impact TBI vs. blast TBI vs. ECI) on selected indices of brain structure and function at baseline and at the 6-month follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Connie C. Duncan, PhD, Principal Investigator — Center for the Study of Traumatic Stress, Department of Psychiatry, Uniformed Services University of the Health Sciences
Locations (2):
- United States (2):
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Fort Belvoir Community Hospital, Fort Belvoir, Virginia

IPD SHARING:
Plan to Share IPD: Yes